CLINICAL TRIAL: NCT06547606
Title: The Effect of Resistive Inspiratory Muscle Training on Optimizing Lung Function in Individuals With Spinal Cord Injury
Brief Title: Effect of Resistive Inspiratory Muscle Training Optimizing Lung Function in Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dhaka (Other)
Responsible Party: Principal Investigator, Dolan Chapa Lucky, Principal Investigator, University of Dhaka
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRP-BHPI/IRB/07/2024/900
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injury (SCI), Respiratory Complication
Keywords: SCI, Respiratory complication, Lung Function, RIMT, Conventional Physiotherapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This study is a double-blinded randomized controlled trial (RCT), where both participants and assessors were blinded. Participants were randomly allocated to either the experimental group, receiving resistive inspiratory muscle training, or the control group, receiving usual care, allocated using a lottery method.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were allocated to either the intervention group or the control group using a concealed lottery method. Assessors were blinded to the treatments received by participants, ensuring impartial evaluation of outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistive Inspiratory Muscle Training (Experimental): Participants in this group will perform resistive inspiratory muscle training, designed to strengthen respiratory muscles and improve lung function. Training involves inhaling through a device that provides resistance, performed five days a week for four weeks.
  Interventions: Other: Usual Care
- Usual Care (Active Comparator): Participants in this group will receive conservative respiratory physiotherapy, which includes standard techniques aimed at maintaining respiratory function and managing symptoms.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Participants in the control group will recieve usual care.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of resistive inspiratory muscle training (RIMT) in optimizing lung function in individuals with spinal cord injury (SCI). It will also learn about the safety and impact of RIMT on health-related quality of life in this population. The main questions it aims to answer are:

Does RIMT improve respiratory function in individuals with SCI? What impact does RIMT have on the health-related quality of life of participants? What are the perceived exertion or dyspnoea levels in participants undergoing RIMT? Researchers will compare RIMT to conventional respiratory physiotherapy to see if RIMT works to enhance lung function and improve overall respiratory outcomes in individuals with SCI.

Participants will:

Perform resistive inspiratory muscle training along with conventional respiratory physiotherapy 5 days a week for 4 weeks.

DETAILED DESCRIPTION:
Globally, over 15 million people are living with spinal cord injury (SCI), according to the World Health Organization (WHO) in 2024. SCI disrupts the normal functioning of the spinal cord, leading to significant physical and neurological impairments. One of the major challenges in SCI management is respiratory complications, which contribute significantly to morbidity and mortality. Resistive inspiratory muscle training (RIMT) has emerged as a promising intervention to enhance respiratory muscle strength and function, potentially reducing respiratory complications in SCI.

The primary objective of this clinical trial is to evaluate the effectiveness of RIMT in optimizing lung function in individuals with SCI. The study also aims to assess the safety of RIMT and its impact on the health-related quality of life of participants.

Researchers will compare RIMT to conventional respiratory physiotherapy to see if RIMT works to enhance lung function and improve overall respiratory outcomes in individuals with SCI.

The study population will consist of individuals with cervical spinal cord injury (SCI) who have impaired respiratory function and are admitted for inpatient rehabilitation. The inclusion criteria include individuals aged 18 to 65 years with cervical cord injury and impaired respiratory function. Exclusion criteria include progressive diseases, head injury, psychiatric conditions, medical instability, ventilator dependency, and the presence of a tracheostomy.

The clinical trial will be conducted at the Spinal Cord Injury Unit of the Centre for the Rehabilitation of the Paralyzed (CRP) in Savar, Dhaka. The CRP provides comprehensive rehabilitation services to patients from all over Bangladesh, ensuring that the study population reflects a broad demographic and economic spectrum.

This study is designed as a randomized controlled trial (RCT) with participants randomly allocated to either the intervention group or the control group. The intervention group will receive resistive inspiratory muscle training (RIMT) in addition to conventional respiratory physiotherapy, while the control group will receive only conventional respiratory physiotherapy.

Data collection will involve a range of tools to assess primary and secondary outcomes:

1. Incentive Spirometry: Assesses lung function.
2. Peak Flow Meter: Measures Peak Expiratory Flow (PEF), assessing expiratory flow rate during forced expiration.
3. SF-12 Health Survey: Assesses health-related quality of life (HRQoL) across various physical and mental health aspects.
4. Modified Borg Scale: Subjective assessment of perceived exertion and dyspnoea.
5. Structured Questionnaire: To gather socio-demographic indicators and additional relevant data.

Data will be analyzed using SPSS version 22. Descriptive statistics will include pie charts, bar charts, and linear line diagrams. Parametric tests such as paired t-tests and unrelated t-tests will be employed to analyze the data. Variables such as mean, mean difference, standard deviations, standard error, degree of freedom, and significance level will be calculated to demonstrate significant differences within and between the experimental and control groups.

By conducting this trial, the study aims to provide robust evidence on the potential benefits of RIMT in improving respiratory function and overall quality of life in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* People with Traumatic Cervical Cord Injury
* Impaired respiratory function

Exclusion Criteria:

* Participants who have Progressive diseases, Head injury, A psychiatric condition , Medical instability, Ventilator dependency, and Presence of tracheostomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Lung function | at baseline and after 4 week
  The spirometer is a medical device used to measure lung function by assessing the volume of air inhaled and exhaled. During a spirometry test, the patient breathes into a mouthpiece connected to the spirometer, which records the amount and rate of air breathed in and out. Key measurements include forced vital capacity (FVC) and forced expiratory volume in one second (FEV1).
Expiratory flow rate during forced expiration | at baseline and after 4 week
  The peak flow meter is a device used to measure how well air moves out of the lungs. It helps assess the peak expiratory flow rate (PEFR), which is the fastest rate at which a person can blow air out of their lungs after taking a deep breath.
Health-Related Quality of Life (HRQoL) | at baseline and after 4 week
  The SF-12 is a validated and reliable health survey that measures health-related quality of life. It comprises 12 questions covering eight domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Responses are used to calculate summary scores for physical and mental health.
Perceived exertion and dyspnoea | at baseline and after 4 week
  The Modified Borg Scale is a validated tool for measuring perceived exertion during physical activity, ranging from 0 (no exertion) to 10 (maximal exertion). It allows individuals to rate their effort intensity, serving as a subjective measure of physical strain.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Mohammad Anwar Hossain, PhD, Study Chair — Professor & Head of Department of Physiotherapy

IPD SHARING:
Plan to Share IPD: No
Participants' demographic details, such as their names and contact information, will be kept confidential by the primary investigator until the publication of the study results. After publication, this information will be discarded.

REFERENCES:
- [Background] Gee CM, Williams AM, Sheel AW, Eves ND, West CR. Respiratory muscle training in athletes with cervical spinal cord injury: effects on cardiopulmonary function and exercise capacity. J Physiol. 2019 Jul;597(14):3673-3685. doi: 10.1113/JP277943. Epub 2019 Jun 11. PMID 31115056
- [Background] McDonald T, Stiller K. Inspiratory muscle training is feasible and safe for patients with acute spinal cord injury. J Spinal Cord Med. 2019 Mar;42(2):220-227. doi: 10.1080/10790268.2018.1432307. Epub 2018 Feb 5. PMID 29400990
- [Background] de Araujo Morais L, Cipriano G Jr, Martins WR, Chiappa GR, Formiga MF, Cipriano GFB. Inspiratory muscle training on quality of life in individuals with spinal cord injury: A systematic review and meta-analysis. Spinal Cord. 2023 Jul;61(7):359-367. doi: 10.1038/s41393-023-00906-1. Epub 2023 Jul 1. PMID 37393409
- [Result] Palermo AE, Butler JE, Boswell-Ruys CL. Comparison of two inspiratory muscle training protocols in people with spinal cord injury: a secondary analysis. Spinal Cord Ser Cases. 2023 Aug 12;9(1):42. doi: 10.1038/s41394-023-00594-2. PMID 37573384
- [Result] Postma K, Haisma JA, Hopman MT, Bergen MP, Stam HJ, Bussmann JB. Resistive inspiratory muscle training in people with spinal cord injury during inpatient rehabilitation: a randomized controlled trial. Phys Ther. 2014 Dec;94(12):1709-19. doi: 10.2522/ptj.20140079. Epub 2014 Jul 31. PMID 25082923
- [Result] Palermo AE, Cahalin LP, Nash MS. A case for inspiratory muscle training in SCI: potential role as a preventative tool in infectious respiratory diseases like COVID-19. Spinal Cord Ser Cases. 2020 Sep 17;6(1):87. doi: 10.1038/s41394-020-00337-7. PMID 32943611